CLINICAL TRIAL: NCT02551419
Title: Effect of a Ketogenic Supplement on Brain Energy Metabolism Measured by Neuroimaging in Mild Cognitive Impairment
Brief Title: Proof of Mechanism of a New Ketogenic Supplement Using Dual Tracer PET (Positron Emission Tomography)
Acronym: BENEFIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2015-509
Record Dates: First submitted 2015-09-15; First posted 2015-09-16 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2019-11

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment; ketones; medium chain triglycerides; Positron emission tomography; magnetic resonance imaging; cognition; brain; neuroimaging
MeSH Terms: conditions — Cognitive Dysfunction; Ketosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ketogenic drink (Experimental): MCT ketogenic drink: ketogenic drink providing 30 g/d of MCT oil in 250 ml of lactose-free skim milk for 6 months supplementation
  Interventions: Dietary Supplement: ketogenic drink
- Placebo (Placebo Comparator): Lactose-free skim milk-based placebo drink containing high-oleic sunflower oil of equivalent energy value to the active arm for a 6 months supplementation
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: ketogenic drink — 6 months' supplementation with the ketogenic drink . Product will be taken daily - 125 ml will be consumed at the morning meal, and 125 ml at the evening meal.
  Arms: ketogenic drink
Dietary Supplement: placebo — 6 months' supplementation with the placebo drink . Product will be taken daily - 125 ml will be consumed at the morning meal, and 125 ml at the
  Arms: Placebo

SUMMARY:
A six month, placebo-controlled, parallel group project in which MCI participants will receive 30 g/day of a custom-made MCT-based ketogenic supplement or a matching placebo. Uptake of both the brain's fuels - ketones (as 11C-AcAc) and glucose (as FDG) - both before and after the intervention will be assessed by PET (position emission tomography) ; imaging and ketone pharmacokinetic as primary objective as well as fMRI, diffusion MRI and cognition.

ELIGIBILITY:
Inclusion Criteria:

* subjective memory complaint
* Montreal Cognitive Assessment (MoCA) score of 18-26/30 or a Mini-mental state exam (MMSE) score of 24-27/30
* autonomy for activity of daily living
* absence of depression

Exclusion Criteria:

* diagnosis of a major cognitive disorder
* diseases or psychiatric disorders that could interfere with participation
* uncontrolled diabetes (fasting plasma glucose >7 mM or glycated hemoglobin >6.5%)
* major depression or history of alcohol or substance abuse within the past 2 years,
* already supplementing with coconut oil or MCT
* vitamin B12 deficiency
* uncontrolled hypertension, dyslipidemia, or thyroid disease,
* visual or hearing impairment impeding comprehension
* participation in another intervention trial
* inability to lie down without moving for 60 min (for the brain imaging)
* presence of implanted metal objects or devices contraindicated for MRI (phase 1)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in global ketone (11C-AcAc) uptake in grey matter | Baseline and 6 months of intervention
  The change in brain ketone uptake will be quantified by PET and expressed as cerebral metabolic rate of AcAc (CMR-A)
Change in plasma ketone | Baseline and 6 months of intervention
  The change in plasma ketone will be measure to obtain a ketone chronic response

SECONDARY OUTCOMES:
Change in global brain FDG uptake in grey matter (CMR-G) | Baseline and 6 months of intervention
  The change in brain glucose uptake will be quantified by PET and expressed as cerebral metabolic rate of glucose (CMR-G)
Change in regional CMR-A | Baseline and 6 months of intervention
  The change in brain ketone uptake will be quantified by PET in different regions of the brain
regional brain volumes by vMRI | Baseline and 6 months of intervention
  Change in brain volume measure by MRI
Change in cognitive status - episodic memory | Baseline and 6 months of intervention
  Change in episodic memory assessed by the 16-item free/cued word learning (Buschke and Grober test- Z score of trial 1, 2, 3 and delay) and the Brief Visuospatial Memory Test-revised (Z score of trial 1)
Change in cognitive status- language domain | Baseline and 6 months of intervention
  Change in language assessed by Boston Naming Test (Z score)
Change in cognitive status - executive function | Baseline and 6 months of intervention
  Change in executive function assessed by condition 4 of the trail making test, condition 3 and 4 of the Stroop test and the 4 conditions of verbal fluency test (all Z score)
Change in cognitive status - processing speed | Baseline and 6 months of intervention
  Change in processing speed assessed by global score of Digit Span (WAIS III), Digit Symbol (WAIS III), condition 1 and 2 of Stroop test and condition 1,2,3,5 of the trail making test (all Z score)
Blood metabolite profile triglycerides | Baseline and 6 months of intervention
  Changes in Triglycerides (mM)
Blood metabolite profile Glucose | Baseline and 6 months of intervention
  Changes in Glucose (mM)
Blood metabolite profile cholesterol | Baseline and 6 months of intervention
  Changes in Total cholesterol (mM)
Derived cerebral metabolic rate of total ketones | Baseline and 6 months of intervention
  Cerebral metabolic rate of total ketone derived from ketone PET (dCMRket, μmol/100 g/min)
Pharmacokinetic ketone response (phase 2) | Baseline and 6 months of intervention
  Area under the curve of pharmacokinetic of blood ketone

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Cunnane, Ph.D., Principal Investigator — Université de Sherbrooke
Locations (1):
- Research Center on Aging, Sherbrooke, Quebec, Canada

REFERENCES:
- [Background] Castellano CA, Nugent S, Paquet N, Tremblay S, Bocti C, Lacombe G, Imbeault H, Turcotte E, Fulop T, Cunnane SC. Lower brain 18F-fluorodeoxyglucose uptake but normal 11C-acetoacetate metabolism in mild Alzheimer's disease dementia. J Alzheimers Dis. 2015;43(4):1343-53. doi: 10.3233/JAD-141074. PMID 25147107
- [Background] Nugent S, Castellano CA, Goffaux P, Whittingstall K, Lepage M, Paquet N, Bocti C, Fulop T, Cunnane SC. Glucose hypometabolism is highly localized, but lower cortical thickness and brain atrophy are widespread in cognitively normal older adults. Am J Physiol Endocrinol Metab. 2014 Jun 1;306(11):E1315-21. doi: 10.1152/ajpendo.00067.2014. Epub 2014 Apr 15. PMID 24735889
- [Background] Nugent S, Tremblay S, Chen KW, Ayutyanont N, Roontiva A, Castellano CA, Fortier M, Roy M, Courchesne-Loyer A, Bocti C, Lepage M, Turcotte E, Fulop T, Reiman EM, Cunnane SC. Brain glucose and acetoacetate metabolism: a comparison of young and older adults. Neurobiol Aging. 2014 Jun;35(6):1386-95. doi: 10.1016/j.neurobiolaging.2013.11.027. Epub 2013 Dec 1. PMID 24388785
- [Background] Courchesne-Loyer A, Fortier M, Tremblay-Mercier J, Chouinard-Watkins R, Roy M, Nugent S, Castellano CA, Cunnane SC. Stimulation of mild, sustained ketonemia by medium-chain triacylglycerols in healthy humans: estimated potential contribution to brain energy metabolism. Nutrition. 2013 Apr;29(4):635-40. doi: 10.1016/j.nut.2012.09.009. Epub 2012 Dec 28. PMID 23274095
- [Background] Cunnane S, Nugent S, Roy M, Courchesne-Loyer A, Croteau E, Tremblay S, Castellano A, Pifferi F, Bocti C, Paquet N, Begdouri H, Bentourkia M, Turcotte E, Allard M, Barberger-Gateau P, Fulop T, Rapoport SI. Brain fuel metabolism, aging, and Alzheimer's disease. Nutrition. 2011 Jan;27(1):3-20. doi: 10.1016/j.nut.2010.07.021. Epub 2010 Oct 29. PMID 21035308

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-11-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT02551419/SAP_000.pdf